CLINICAL TRIAL: NCT00987857
Title: Barrett's Oesophagus Two Yearly Surveillance Versus Endoscopy at Need: a Randomised Controlled Trial to Estimate Effectiveness and Cost-effectiveness Study (BOSS)
Brief Title: Endoscopy Every 2 Years or Only as Needed in Monitoring Patients With Barrett Esophagus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Gloucestershire Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Clive Stokes, Professor Hugh Barr, Gloucestershire Hospitals NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: NHS-GRH-HTA-05/12/01; CDR0000649890 (Registry Identifier: PDQ (Physician Data Query)); ISRCTN54190466
Record Dates: First submitted 2009-09-30; First posted 2009-10-01 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Esophageal Cancer; Precancerous Condition
Keywords: esophageal cancer; adenocarcinoma of the esophagus; Barrett esophagus
MeSH Terms: conditions — Esophageal Neoplasms; Precancerous Conditions; Adenocarcinoma Of Esophagus; Barrett Esophagus | interventions — Endoscopic Mucosal Resection; Endoscopy; High-Throughput Screening Assays

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 yearly endoscopies (Active Comparator): Two years endoscopies
  Interventions: Procedure: 2 yearly endoscopy; Procedure: comparison of screening methods; Procedure: diagnostic endoscopic procedure; Procedure: endoscopic biopsy; Procedure: endoscopic procedure; Procedure: quality-of-life assessment; Procedure: screening method
- endoscopy at need (Experimental): Endoscopy only when patient reports symptoms
  Interventions: Procedure: 2 yearly endoscopy; Procedure: comparison of screening methods; Procedure: diagnostic endoscopic procedure; Procedure: endoscopic biopsy; Procedure: endoscopic procedure; Procedure: quality-of-life assessment; Procedure: screening method

INTERVENTIONS:
Procedure: 2 yearly endoscopy — 2 yearly endoscopy versus endoscopy at need
Procedure: comparison of screening methods — 2 yearly endoscopy versus endoscopy at need
Procedure: diagnostic endoscopic procedure — 2 yearly endoscopy versus endoscopy at need
Procedure: endoscopic biopsy — 2 yearly endoscopy versus endoscopy at need
Procedure: endoscopic procedure — 2 yearly endoscopy versus endoscopy at need
Procedure: quality-of-life assessment — QOL aims to elicit any differences in QOL between 2 yearly endoscopy versus endoscopy at need
Procedure: screening method — All Barretts patients to be screened

SUMMARY:
RATIONALE: Screening tests may help doctors find cancer cells early and plan better treatment. It is not yet known whether endoscopy every 2 years is more effective than endoscopy only as needed in finding esophageal cancer in patients with Barrett esophagus.

PURPOSE: This randomized phase III trial is studying endoscopy every 2 years to see how well it works compared with endoscopy only as needed in monitoring patients with Barrett esophagus.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To establish whether endoscopic surveillance every 2 years or endoscopy at need only is superior in terms of overall survival and, if neither is superior, whether endoscopy at need only is non-inferior to surveillance every 2 years in patients with Barrett esophagus.

Secondary

* To estimate the cost-effectiveness of endoscopic surveillance every 2 years as compared to endoscopy at need only.
* To establish whether there is a significant difference between endoscopic surveillance every 2 years or endoscopy at need only in terms of the incidence of esophageal cancer, gastric or esophageal cancer, or all cancers.
* To establish whether there is a significant difference between endoscopic surveillance every 2 years or endoscopy at need only in terms of the time to diagnosis of esophageal adenocarcinoma.
* To establish whether there is a significant difference between endoscopic surveillance every 2 years or endoscopy at need only in terms of the stage of esophageal adenocarcinoma at diagnosis using TNM staging.
* To establish whether there is a significant difference between endoscopic surveillance every 2 years or endoscopy at need only in terms of morbidity and mortality related to endoscopy, esophageal surgery, and other endoscopy-related interventions (e.g., ablation).
* To establish whether there is a significant difference between endoscopic surveillance every 2 years or endoscopy at need only in terms of the frequency of endoscopy.

OUTLINE: This is a multicenter study. Patients are stratified according to age at diagnosis (< 65 years vs ≥ 65 years), length of Barrett metaplasia segment including tongues (< 2 cm vs ≥ 2 cm and ≤ 3 cm vs > 3 cm and ≤ 8 cm vs > 8 cm), and newly diagnosed disease (defined as the date of endoscopy confirming Barrett metaplasia was within the past 4 months) (yes vs no). Patients are randomized to 1 of 2 intervention arms.

* Arm I: Patients undergo surveillance endoscopy with quadrantic biopsies taken every 2 cm. Patients undergo endoscopy every 2 years for a total of 6 endoscopies over 10 years.
* Arm II: Patients undergo endoscopy as needed over 10 years. All patients may undergo urgent endoscopy if they develop dysphagia, unexplained weight loss of > 7 lb, iron-deficiency anemia, recurrent vomiting, or worsening upper gastrointestinal symptoms.

All patients complete a questionnaire that includes a quality-of-life measure and questions about medication at baseline, every 2 years, and following key events (e.g., diagnosis of any cancer or high-grade dysplasia).

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed circumferential Barrett metaplasia meeting 1 of the following criteria:

  * At least 1 cm from the gastro-esophageal junction
  * At least a 2 cm non-circumferential tongue of Barrett metaplasia
* Undergone endoscopy within the last 2 years to confirm Barrett metaplasia and exclude high-grade dysplasia and carcinoma
* No known high-grade dysplasia or carcinoma

PATIENT CHARACTERISTICS:

* Resident of the United Kingdom
* Informed of the risk of Barrett esophagus developing into esophageal cancer, either at the visit when the invitation letter is issued or on a documented previous occasion
* Able to undergo endoscopy
* No medical conditions that would make endoscopy difficult or hazardous

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3400 (Actual)
Dates: Start 2009-03; Primary Completion 2022-05 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Overall survival

SECONDARY OUTCOMES:
Cost-effectiveness
Incidence of esophageal cancer, gastric or esophageal cancer, or all cancers
Time to diagnosis of esophageal adenocarcinoma
Stage of esophageal adenocarcinoma at diagnosis using TNM staging
Morbidity and mortality related to endoscopy, esophageal surgery, and other endoscopy-related interventions
Frequency of endoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Hugh Barr, Principal Investigator — Gloucestershire Hospitals NHS Foundation Trust
Locations (1):
- Gloucestershire Royal Hospital, Gloucester, England, United Kingdom

REFERENCES:
- [Derived] Old O, Jankowski J, Attwood S, Stokes C, Kendall C, Rasdell C, Zimmermann A, Massa MS, Love S, Sanders S, Deidda M, Briggs A, Hapeshi J, Foy C, Moayyedi P, Barr H; BOSS Trial Team. Barrett's Oesophagus Surveillance Versus Endoscopy at Need Study (BOSS): A Randomized Controlled Trial. Gastroenterology. 2025 Nov;169(6):1233-1243.e8. doi: 10.1053/j.gastro.2025.03.021. Epub 2025 Apr 1. PMID 40180292